CLINICAL TRIAL: NCT02418715
Title: Effects of Water-Based Exercise on Lipid Profile and Lipoprotein Lipase of Dyslipidemic Premenopausal Women: A Randomized Controlled Trial
Brief Title: Effects of Water-Based Exercise on Lipid Profile and Lipoprotein Lipase of Dyslipidemic Premenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Rochelle Rocha Costa, MSC, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Water-Based Exercise Trial
Record Dates: First submitted 2015-04-08; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Water Aerobics Training (Experimental): The training period was composed by a 12-week macrocycle with two sessions per week. The macrocycle was divided into three four-week mesocycles that were, in turn, divided into four one-week microcycles composed by two training sessions. Each training session took 45 min. Nine different water-aerobics exercises were used during the training period. These exercises were performed alternating the right and left limbs. Exercise intensities were controlled using the Borg Scale. Interval training was used alternating intensities ranged between 9 (easy) and 15 (hard). During the first mesocycle, participants performed sets of 3min at intensity 13 interspersed by 2min at intensity 9; during the second mesocycle, sets of 3min at intensity 15 followed by 2min at intensity 9 were performed; finally, sessions of the third mesocycle were composed by sets of 3min at intensity 15 followed by 2min at intensity 11.
  Interventions: Other: Water Aerobics Training
- Control (No Intervention): No training, no intervention.

INTERVENTIONS:
Other: Water Aerobics Training
  Other Names: HA
  Arms: Water Aerobics Training

SUMMARY:
The aim of this study was to investigate the effects of water-based exercises on lipid profile (LP) and lipoprotein lipase (LPL) levels in premenopausal dyslipidemic women.

It was hypothesized that a water-based aerobic interval-training period would decrease plasma concentrations of atherogenic lipoproteins and concomitantly increase HDL and LPL levels, as well as maximal oxygen uptake (VO2max) values.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Sedentary
* Dyslipidemic
* Aged between 40 and 50 years old

Exclusion Criteria:

* Smokers
* Hypolipemic drugs users

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Lipid Profile Levels (total cholesterol, LDL, HDL, triglycerides) | 12 weeks

SECONDARY OUTCOMES:
Lipoprotein Lipase Levels | 12 weeks

OTHER OUTCOMES:
Maximal oxygen uptake (VO2max) values | 12 weeks